CLINICAL TRIAL: NCT02426645
Title: Microcirculatory Alteration and Biomarkers: New Approach for Early Assessment of Septic Multi-organ Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Prof. Dr. Marc-H. Dahlke, Ph. D. (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Marc-H. Dahlke, Ph. D., Professor, University Hospital Regensburg
Organization: University Hospital Regensburg (Other)
Other Study IDs: Mibisep
Record Dates: First submitted 2015-04-16; First posted 2015-04-27 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Sepsis; Multiple Organ Failure
Keywords: Biomarkers; Sepsis; Multi organ dysfunction; Immunomonitoring; CEUS
MeSH Terms: conditions — Sepsis; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to investigate associations between early structural cellular injury and microvascular alteration with progression of septic organ dysfunction according to total SOFA-Score (an ICU-scoring system - the Sequential Organ Failure Assessment Score). Patients will be monitored for renal (TIMP-2, IGFBP7), and intestinal biomarkers (plasma i-FABP) in conjunction with kidney and muscle vascular bed microvascular perfusion analysis assessed by contrast-enhanced ultrasonography (CEUS). In parallel, a comprehensive analysis of patients' immunological status will be conducted using an established, on-site immune monitoring panel.

The ultimate goal of this study is an early identification of septic patients developing multiorgan dysfunction which may facilitate a timely novel intervention in the future to improve outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients ≥18 years of age with severe sepsis and fulfill the following criteria at the admission to ICU:

* Peritonitis (abdominal infection) and performed source control (either surgically or interventionally)
* 2 or more criteria for systemic inflammatory response syndrome (temperature >38° or<36°; heart rate >90 beats per minute; respiratory rate >20 breaths per minute or paCO2 <32 mmHg; white blood cell count >12,000/mm3, <4000mm3 or >10% immature forms) and serum lactate level of 4mmol/l and more or refractory hypotension - mean arterial pressure <65mmHg or systolic blood pressure <90mmHg after fluid challenge of 1000ml or more /30min
* Absence of any familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Written informed consent prior to any study procedures

Exclusion Criteria:

* Pre-existing renal-replacement therapy in the pre-operative course
* Pre-existing shock
* Acute coronary syndrome
* Active hemorrhage
* Trauma
* Known allergy to ultrasound contrast media
* Anemia with hemoglobin concentration < 7g/dl
* Patients not able to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with severe sepsis of abdominal origin within 24h after onset and performed source control
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-01 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of early post-operative course of novel cellular injury biomarkers as well as microvascular perfusion in critically ill patients with severe sepsis and to collection any first evidence of the association of these markers with the SOFA-Score | 60 weeks

SECONDARY OUTCOMES:
28 day mortality | 60 weeks
90 day mortality | 60 weeks
Length of ICU stay | 60 weeks
Length of hospital stay | 60 weeks
Early post-operative course of microvascular perfusion of the kidney and muscle vasculature bed using CEUS | 60 weeks
Incidence of acute kidney injury (AKI) within the first 48 hours as based on current Kidney Disease: Improving Global Outcomes (KDIGO) recommendation | 60 weeks
Incidence of acute kidney injury (AKI) within the first 7 days as based on current Kidney Disease: Improving Global Outcomes (KDIGO) recommendation | 60 weeks
Need for renal replacement therapy (RRT) after admission to ICU | 60 weeks
Identification of an "immunological fingerprint" indicating multi-organ dysfunction | 60 weeks
  Flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Marc H Dahlke, Prof. Dr., Principal Investigator — University Hospital Regensburg
Locations (1):
- Department of Surgery, University Hospital Regensburg, Regensburg, Bavaria, Germany